CLINICAL TRIAL: NCT03551860
Title: A Comparative Evaluation of Quadratus Lumborum Block Versus Fascia Iliaca Nerve Block for Patients Undergoing Elective Total Hip Replacement Under Spinal Anaesthesia
Brief Title: Quadratus Lumborum Block Versus Fascia Iliaca Nerve Block for Patients Undergoing Total Hip Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Adelaide and Meath Hospital, incorporating The National Children's Hospital (Other)
Responsible Party: Principal Investigator, Karthikeyan Kallidaikurichi Srinivasan, Consultant Anaesthetist, The Adelaide and Meath Hospital, incorporating The National Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017/1/01-2018-01
Record Dates: First submitted 2018-03-23; First posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Hip Replacement
Keywords: Total hip replacement; Motor block post-operatively; Morphine consumption post-operatively; Transmuscular Quadratus Nerve Block; Fascia Iliaca Nerve Block

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to nature of intervention (one single injection vs a second single injection in different anatomical location) the participant and the care provider cannot be blinded.The investigator will use an already filled data collection sheet and enter randomised data into a master file. The data will be analysed by an individual blinded to the which group the participant was in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQL Group (Experimental): Administration of a single shot transmuscular quadratus lumborum (TQL) peripheral nerve block following spinal neuraxial blockade.
  Interventions: Procedure: TQL
- FIB Group (Active Comparator): Administration of a single shot fascia iliac (FIB) peripheral nerve block following spinal neuraxial blockade.
  Interventions: Procedure: FIB

INTERVENTIONS:
Procedure: TQL — For the intervention of TQL peripheral nerve block the needle tip will be advanced by in-plane technique and local anaesthetic will be deposited between psoas major and quadratus lumborum muscles. 20 ml of 0.25% bupivacaine will be administered under ultrasound guidance following careful intermittent aspiration. The needle tip will not be repositioned unless the patient complains of paraesthesia.
  For the intervention of spinal neuraxial blockade the needle will be advanced into the subarachnoid space. Once clear CSF is visualised 3.2ml 0.5% plain bupivacaine will be infiltrated.
  Other Names: Transmuscular Quadratus Nerve Block
  Arms: TQL Group
Procedure: FIB — The needle tip will be advanced by in-plane technique and local anaesthetic will be deposited deep to the fascia iliaca. 20ml of 0.25% bupivacaine will be administered under ultrasound guidance following careful intermittent aspiration. The needle tip will not be repositioned unless the patient complains of paraesthesia.
  For the intervention of spinal neuraxial blockade the needle will be advanced into the subarachnoid space. Once clear CSF is visualised 3.2ml 0.5% plain bupivacaine will be infiltrated.
  Other Names: Fascia Iliaca Nerve Block
  Arms: FIB Group

SUMMARY:
Investigators hypothesise that for patients undergoing elective total hip replacements, a single injection Transmuscular Quadratus Lumborum (TQL) block, when compared to a single injection Fascia Iliaca Block (FIB), will provide better analgesia and less motor block in the initial 24 hour period.

DETAILED DESCRIPTION:
Total hip replacement is a commonly performed surgical procedure with up to 4,500 procedures performed annually in Ireland and up to 400,000 per year in the United States. Most of the patients experience moderate to severe pain in the initial post-operative period. Multimodal analgesia with peripheral nerve blockade is recommended as the gold standard modality for management of lower limb joint replacements. The limitations with peripheral nerve block include duration of therapy with single shot injections and associated motor block which can delay rehabilitation.

Transmuscular Quadratus Lumborum injection has been described recently as an effective option for post-operative analgesia in patients undergoing total hip replacement. Single injection can provide analgesia for up to 24 hours. We aim to investigate if a TQL block when compared to FIB provides superior analgesia and less motor block in the acute post-operative period.

All patients scheduled for elective hip replacement surgery will be contacted prior to the surgery (at least 24 hours) over the telephone and information about the nature and purpose of the study will be provided to them by Anaesthesia personnel who are involved in the study. They will be directed to a dedicated page on our website to further inform themselves, if desired. Written informed consent will be obtained from all patients prior to participation in the study. Patients can remove their consent without question at any time during or after the study.

Patients will be randomised to either the TQL group (intervention group) or FIB group (conventional group) by computer generated random numbers and allocation will be enclosed in sealed envelopes. Due to the nature of the intervention, the Anaesthetist performing/supervising the block and patient receiving the block cannot be blinded. Outcome measurements will be recorded by study observers blinded to the group allocation.

On arrival to the Anaesthesia induction room baseline monitoring (non-invasive blood pressure, pulse oximetry and 3-lead ECG) and intravenous access will be established. Patients in both groups will be positioned sitting on a level trolley with feet resting on a foot rest. They will be given a pillow to hug and requested to maintain an arched back posture with an assistant holding the patient to aid positioning. No sedation will be given prior to or during administration of spinal anesthesia.

Spinal anaesthesia will be performed under strict aseptic precautions (Chlorhexidine 0.5% for skin decontamination with anaesthetist performing the procedure scrubbed wearing sterile gown, cap and sterile gloves). A 25G Whitacre needle will be used and 3.2ml 0.5% plain bupivacaine will be infiltrated into the intrathecal space.

Transmuscular Quadratus Lumborum Block (TQL):

Following the administration of spinal anaesthetic, the patient will be positioned laterally with the operating side as the non dependant side. Skin decontamination of the block site will be carried out with 2% Chlorhexidine (Chloraprep 3 ml applicator, CareFusion Corporation, San Diego, CA 92130,USA). Under strict aseptic precautions (cap, mask, sterile gloves, sterile probe cover and sterile ultrasound gel), a 100 mm (Stimuplex® Ultra 360® 22 gauge insulated echogenic needle with 30° bevel and extension set) needle will be used to perform TQL block. A curvilinear low frequency probe (2-5 MHz) will be placed above the iliac crest and the following structures will be identified i) Transverse process ii) Erector spinae muscle iii) Quadratus lumborum muscle iv) Psoas major muscle. The needle will be advanced by in-plane technique and local anaesthetic will be deposited between psoas major and quadratus lumborum muscles. 20 ml of 0.25% bupivacaine will be administered under ultrasound guidance following careful intermittent aspiration.

Fascia Iliaca Block (FIB):

Following the administration of spinal anaesthetic, the patient will be positioned supine. Skin decontamination of the block site will be carried out with 2% Chlorhexidine (Chloraprep 3 ml applicator, CareFusion Corporation, San Diego, CA 92130,USA). Under strict aseptic precautions (cap, mask, sterile gloves, sterile probe cover and sterile ultrasound gel), an 80 mm (Stimuplex® Ultra 360® 22 gauge insulated echogenic needle with 30° bevel and extension set) needle will be used to perform FIB. A linear high frequency probe (8-13 MHz) will be placed along the inguinal crease to identify the femoral artery, femoral nerve and Iliacus fascia. The needle will be advanced by in-plane technique and local anaesthetic will be deposited under the fascial iliaca. 20 ml of 0.25% bupivacaine will be administered under ultrasound guidance following careful intermittent aspiration.

All patients (unless contraindicated) will receive intra-operative intravenous medication as follows: paracetamol 1g, Parecoxib 40mg, tranexamic acid 1g and antibiotics as per local guidelines. Perioperative sedation will be left to the discretion of the anaesthetist. Following transfer to the recovery unit if patient reports pain score by numerical rating score (NRS) > 3, morphine 2 mg increments will be given intravenously by the recovery staff. This will be repeated every 5 minutes till the pain score is <4. In patients requiring more than 10 mg of morphine in the recovery, an Anaesthetist will be requested to review the patient. Post-operatively, in the absence of contraindications, all patients will be prescribed regular Paracetamol 1g every 6 hours and Celecoxib 200 mg every 12 hours. Anti-emetics (Ondansetron 4 mg every 8 hours and Cyclizine 50 mg every 8 hours) will be prescribed for all patients to be administered as required. All patients will receive morphine PCA in the post-operative period. All patients will be reviewed at 6 hours and 24 hours post peripheral nerve block insertion to assess their pain scores (NRS) and motor block.

Statistics:

A sample size of 46 patients (23 per group) is estimated based on 50% reduction in morphine consumption with power of 80% and alfa error of 0.05%. To allow for drop outs,investigators aim to recruit 50 patients in total.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective total hip replacements under spinal anaesthesia
* ASA 1-3
* Age > 18 yrs.
* Patient is able to provide written informed consent

Exclusion Criteria:

* Local infection
* Allergy to local anaesthetics
* Severe coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-04-10 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
24 hour morphine consumption between the two groups | 24 hour post-operative period
  Intravenous Patient Controlled Analgesia (PCA) Morphine will be set up and explained to all participants. The AMNCH hospital standard will be use. This is 2mg/ml concentration; 1mg dose; 6 minute lockout period between administration; maximum morphine consumption of 40mg within a 4 hour period.

SECONDARY OUTCOMES:
Motor Block | 24 hours post-operative period - measured at 6 and 24 hours
  Modified Bromage Scale for use in Lower Limb will be used to assess residual motor block.
  Scale ranges:
  1. Complete block (unable to move feet or knee)
  2. Almost complete block (able to move feet only)
  3. Partial block (just able to move knees)
  4. Detectable weakness of hip flexion while supine (full flexion of knees)
  5. No detectable weakness of hip flexion while supine
  6. Able to perform partial knee bend.
  The higher the number value the better the outcome is considered to be and the less the residual nerve block.
Numerical Rating Scale (NRS) for Pain | 24 hours post-operative period - measured at 6 and 24 hours
  A Numerical Rating Scale is an 11 point scale that involves asking a patient to rate his or her pain from 0 to 10 with the understanding that 0 is equal to no pain and 10 is equal to the worst pain possible. The patient provides a verbal response to which the assessor can document the intensity of pain the patient reports.

CONTACTS AND LOCATIONS:
Overall Officials: Karthikeyan K Srinivasan, MD.,FCARCSI, Principal Investigator — Adelaide and Meath Hospital, Incorporating National Children's Hospital
Locations (1):
- Adelaide and Meath Hospital, Incorporating National Children Hospital, Tallaght, Dublin 24, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petis SM, Howard JL, Lanting BA, Marsh JD, Vasarhelyi EM. In-Hospital Cost Analysis of Total Hip Arthroplasty: Does Surgical Approach Matter? J Arthroplasty. 2016 Jan;31(1):53-8. doi: 10.1016/j.arth.2015.08.034. Epub 2015 Aug 29. PMID 26387922
- [Background] Gaffney CJ, Pelt CE, Gililland JM, Peters CL. Perioperative Pain Management in Hip and Knee Arthroplasty. Orthop Clin North Am. 2017 Oct;48(4):407-419. doi: 10.1016/j.ocl.2017.05.001. Epub 2017 Jun 29. PMID 28870302
- [Background] Ueshima H, Yoshiyama S, Otake H. RETRACTED: The ultrasound-guided continuous transmuscular quadratus lumborum block is an effective analgesia for total hip arthroplasty. J Clin Anesth. 2016 Jun;31:35. doi: 10.1016/j.jclinane.2015.12.033. Epub 2016 Mar 22. PMID 27185672 (Retraction: PMID 35393191 J Clin Anesth. 2022 Aug;79:110702; PMID 35397960 J Clin Anesth. 2022 Aug;79:110704)
- [Background] La Colla L, Uskova A, Ben-David B. Single-shot Quadratus Lumborum Block for Postoperative Analgesia After Minimally Invasive Hip Arthroplasty: A New Alternative to Continuous Lumbar Plexus Block? Reg Anesth Pain Med. 2017 Jan/Feb;42(1):125-126. doi: 10.1097/AAP.0000000000000523. No abstract available. PMID 27997495

DOCUMENTS (2):
  • Informed Consent Form (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/60/NCT03551860/ICF_000.pdf
  • Study Protocol (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/60/NCT03551860/Prot_001.pdf